CLINICAL TRIAL: NCT05353400
Title: At Home Early vs. Delayed Catheter Removal Following Failed Postoperative Voiding Trial: a Randomized Trial
Acronym: AHEADCARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment and attrition of study personnel
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00083499; V13-30-2022 (Other: AtriumHealth)
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Urinary Retention Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Intervention group): self-removal of transurethral catheter on POD 1 (Experimental): Subjects will self-remove transurethral catheter at home on postop day 1
  Interventions: Other: Early urinary catheter removal
- (Standard practice group): self-removal of transurethral catheter on POD 3 (Active Comparator): Subjects will self-remove transurethral catheter at home on postop day 3
  Interventions: Other: Urinary catheter removal on POD 3

INTERVENTIONS:
Other: Early urinary catheter removal — Early catheter removal
  Other Names: Catheter Removal on POD 1
  Arms: (Intervention group): self-removal of transurethral catheter on POD 1
Other: Urinary catheter removal on POD 3 — Catheter removal on POD 3
  Arms: (Standard practice group): self-removal of transurethral catheter on POD 3

SUMMARY:
This study aims to investigate whether patients who self-remove their indwelling transurethral catheters on POD 1 have similar rates of postoperative catheter reinsertion for urinary retention (within the first 7 days after surgery) compared with those who undergo catheter self-removal on POD 3.

DETAILED DESCRIPTION:
Studies estimate the rate of post-operative urinary retention (POUR) after pelvic reconstructive surgery to be between 2.5-43% in all patients1. Consequently, patients undergoing pelvic reconstructive surgery will commonly undergo an assessment of voiding function prior to discharge. Patients who do not successfully complete a voiding trial (VT) are typically discharged from the hospital with a transurethral indwelling catheter. The preferred length of time the catheter remains in place postoperatively, however, varies widely (1 to 7 days) amongst pelvic reconstructive surgeons2-4.

Over the past few years, Enhanced Recovery After Surgery (ERAS) protocols have been adopted for patients undergoing reconstructive vaginal and minimally invasive (laparoscopic or robotic) surgery with increased focus on patient centered outcomes5. The benefits of ERAS in pelvic reconstructive surgery often allow for patients to be discharged home from the hospital the same day of their surgery. Unfortunately, same day discharge is associated with higher rates of postoperative voiding dysfunction and subsequent discharge home with a urinary catheter, with an incidence reported as high as 33.9-36%2,6. This increased rate of postoperative urinary retention has been reflected in our patient population. Prior to the implementation of ERAS in our pelvic reconstructive surgery division at Atrium Health, the rate of discharge home with a urinary catheter after failed VT on postoperative day (POD) 1 was 28%. With the implementation of an ERAS protocol and same day discharge (POD 0), the rate climbed to 43%7. Consequently, a higher percentage of postoperative patients have required a second VT prior to catheter discontinuation. This has necessitated additional clinical visits with a nurse or other provider, further stretching our clinical staff and obligating patients to make an additional trip to the clinic for a repeat postoperative VT.

Recent evidence supports the safety and improved patient experience in patients who self-discontinue a transurethral urinary catheter. In the study by Shatkin-Margolis et al., patients who had undergone pelvic reconstructive surgery were randomized to either self- discontinuation or in office discontinuation overseen by medical personnel one week after surgery8. This study found that self-discontinuation of transurethral catheter was non-inferior to office-based discontinuation following pelvic reconstructive surgery. Additionally, the authors found that self-discontinuation resulted in fewer patient encounters and improved patient experience.

Given this supportive evidence of safe catheter self-discontinuation and our practice's desire to improve patient satisfaction while decreasing clinical burden, we have adopted a practice where the patient self-removes their urinary catheter on the same day that a typical in-office VT would occur (POD 3). During preoperative counseling visits, our patients receive structured handouts with pictorial and descriptive language explaining how to safely self-remove a transurethral catheter (Figure 1). If VT failure should occur, the post anesthesia care unit (PACU) nursing staff review the instructions once again with the patient and the patient's support person(s) prior to discharge. Patients are told to call the office with any symptoms or concerns. Additionally, a nurse from our practice follows up with the patient via telephone on POD 1.

Patient experience following surgery is an important patient centered outcome. Unfortunately, being discharged home with an indwelling transurethral catheter for any amount of time is often perceived by patients as a postoperative complication and is a source of dissatisfaction in patients undergoing pelvic reconstructive surgery9-10. Therefore, decreasing the dissatisfaction surrounding postoperative catheter use improves the patient experience. Several studies have evaluated early postoperative catheter discontinuation after pelvic reconstructive surgery in an effort to limit the length of time that a catheter is in place. In a randomized controlled trial of immediate versus POD1 catheter removal in patients undergoing minimally invasive pelvic reconstructive surgery by Vallabh-Patel et al. the rate of POUR on POD 0 was 31%; however, the rate on POD 1 was 4.5%2. Similar low rates of POUR were noted in a prospective cohort trial performed by Botros et al. which evaluated the effects of a mid-urethral sling at the time of robotic sacrocolpopexy and noted a POD 1 retention rate of 1% in this patient population11. Finally, in a retrospective cohort study incorporating both laparoscopic and vaginal pelvic reconstructive surgery performed by El Hiraki et al., the rate of failed VT within 23 hours of surgery was 11.1% for minimally invasive group and 34% for the vaginal surgery group12. This limited body of evidence suggests that a voiding trial as early as postoperative day 1 seems to yield a voiding trial pass rate of 1-34% in pelvic reconstructive surgery patients.

Our group aims to optimize urinary catheter management for both the patient and the clinical staff in the postoperative period when patients are discharged on the same day of their surgery with a transurethral urinary catheter. We are proposing a non-inferiority trial comparing at home POD 1 catheter removal with at home POD 3 catheter removal (our current standard of practice).

ELIGIBILITY:
Inclusion Criteria:

* English speaking Age 18+ Undergoing pelvic reconstructive surgery with ERAS protocol Incomplete bladder emptying after same day VT in PACU (as defined by an ultrasound or straight catheter post void residual of greater than 50% the total instilled volume within 10 minutes following a void postoperatively) Able to complete a telephone appointment on either postoperative day 1 or 3

Exclusion Criteria:

* Active urinary tract infection, defined by CDC criteria Patients undergoing pelvic reconstructive surgery where ERAS protocol is not utilized (examples: isolated Labiaplasty, chemodenervation with onabotulinum toxin A, urethral bulking, mid-urethral sling, sacral neuromodulation) Contraindication to ERAS protocol and/or its medications Elevated pre-op PVR greater than 200mL (on urodynamic testing or uroflow or straight catheter sample, that remains elevated after prolapse is reduced) Limited manual dexterity (limiting self-removal of catheter) Intra-op cystotomy or urinary tract injury Planned long term catheterization (e.g., fistula repair, urethral diverticulum) Planned hospital admission or patients who are not discharged from hospital the same day of their surgery Pregnancy Dependent on catheterization to void preoperatively Patients who request clean intermittent catheterization (CIC) after immediate failed VT Neurological conditions that affect voiding function (examples: spinal cord lesions, multiple sclerosis, Parkinson's disease, past stroke history with residual neurologic deficits) Concomitant surgical procedure by another service Conversion to open surgery Patients discharged to nursing home or rehabilitation care facility

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients requiring re-insertion of a transurethral urinary catheter | 7 days
  Percentage of patients with urinary retention requiring re-insertion of a transurethral urinary catheter or needing to do self catheterization within one week of surgery after catheter self-discontinuation on either POD 1 or POD 3 following pelvic reconstructive surgery utilizing ERAS protocol.

SECONDARY OUTCOMES:
Short Term Catheter Burden Questionnaire | 7 days
  Postoperative patient satisfaction using validated questionnaire-Short Term Catheter Burden Questionnaire (STCBQ)13 recorded on day of catheter removal.
  Total scale score from 5 to 30. Higher scores indicate greater embarrassment/bother.
Urinary Force of stream | 7 days
  Urinary Force of stream (FOS) reported in millimeters (mm) on visual analog scale (VAS) for first void after catheter removal 14-15 (Figure 3) recorded on day of catheter removal
Urinary tract infection rate | 30 days
  Urinary tract infection (UTI) rates-first 30 days after surgery defined by the CDC criteria
  This will be reported as an absolute number and calculated and reported as a percentage of the total number of patients who had a UTI/ total number of patients in the study.
Number of patient phone calls | 7 days
  Number of patient phone calls to triage nursing or clinic in first 7 days following surgery
Number of visits | 30 days
  Number of visits (Emergency room/clinic/post anesthesia care unit (PACU), other) for catheter reinsertion within 30 days of surgery
Readmission rates | 30 days
  30-day readmission rates
Prolonged catheterization | 30 days
  Need for prolonged catheterization or clean intermittent self catheterization (CIC) for greater than 7 days
  This will be reported as an absolute number and calculated and reported as a percentage of the total number of patients who required greater than 7 days of catheterization/ total number of patients in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Tarr, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT05353400/ICF_000.pdf